CLINICAL TRIAL: NCT01626274
Title: Long Term Vital Parameter Monitoring Pilot Study to Evaluate Measurement Data Via In-ear Sensor in Comparison to Standard Polysomnography in Sleep Laboratory
Brief Title: Long Term Vital Parameter Monitoring (LAVIMO)
Acronym: LAVIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CTC-A_10-016; EK 231/10 (Other: Ethics Committee University Hospital Aachen)
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Polysomnography; Long term vital signs monitoring; In-ear sensor system; Photoplethysmographic micro-optic device; High wearing comfort
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: in-ear sensor (Experimental): Patients who routinely undergo a polysomnography night (1 night) are monitored via in-ear sensor which will be embedded in the auditory canal. During this night vital signs parameters are monitored, processed and subsequently compared to the polysomnography data.
  Interventions: Device: LAVIMO in- ear sensor system

INTERVENTIONS:
Device: LAVIMO in- ear sensor system — Long term vital signs parameters like heart rate, heart rate variability, breathing and oxygen saturation are measured via in- ear sensor system during 1 polysomnographic night
  Other Names: Photoplethysmographic microoptic reflective microsensor

SUMMARY:
The purpose of this study is to evaluate the feasibility of non-intrusive 24 hours non-invasive measurements with minimized LAVIMO sensor system. The LAVIMO-system is a photoplethysmographic device for reflective mode measurements of the optical damping upper skin layers inside of the ear canal at two different wave lengths. It consists of the in-ear sensor, the electronics and a PC. Vital signs parameter like heart rate, heart rate variability, breathing and arterial blood oxygenation are monitored in patients with sleep apnoea and compared to measurements of standard polysomnography of these patients during one night in the sleep laboratory.

DETAILED DESCRIPTION:
In 20 patients who routinely have to undergo a polysomnographic night in sleep laboratory LAVIMO measurements like heart rate, heart rate variability, breathing and arterial blood oxygenation are performed parallel to standard polysomnography measurements and subsequently compared to the data of the standard polysomnography. The LAVIMO sensor system consists of the in- ear sensor, the electronics and a PC; the individually formed sensor is embedded into an ear mould for proper fit inside the ear canal. Inside two LEDs emit light into the adjacent skin at 760 and 905 nm wavelengths. The intensity of the backscattered light is detected by a photo detector. In the electronics, the control signals for the LEDs are provided, as well as the photo detector signal is further processed and A-D converted. The electronics also provide a wireless connection to the PC via bluetooth. Data recording, post processing and displaying are tasks of the PC. The feasibility of non- intrusive 24 hours and non-invasive measurements like heart rate, heart rate variability, breathing and oxygen saturation is proved via this minimized sensor and electronics placed at a suitable place at the body guaranteeing high wearing comfort. This includes a wireless data communication for unrestricted mobility. Subsequently the data are compared to the standard polysomnography data to extract vital signs or for example to recognize possible phases of sleep apnoea. The goal in future refering to preventive medical monitoring will be early detection of risk factors for patient's health and improvement of living conditions.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years who routinely have to undergo a polysomnography night
* sleep apnoea patient
* able to give informed consent

Exclusion Criteria:

* dementia
* cochlea implant
* severe lung diseases
* allergy against material of the sensor
* inflammation of the middle ear
* inflammation of auditory canal
* occlusion because of cerumen
* electric implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Extraction of vital signs out of measurement data via individually formed in-ear sensor system in comparison to standard polysomnography data in sleep laboratory | one night
  during one polysomnographic night in sleep laboratory the patient will receive the LAVIMO in- ear sensor system and vital parameters like heart rate, heart rate variability, breathing and oxygen saturation will be monitored. Subsequently the data will be processed and compared to the standard polysomnographic data

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schiefer, MD, Principal Investigator — Neurological Clinic, University Hospital Aachen
Locations (1):
- Neurological Clinic , University Hospital, Aachen, North Rhine-Westphalia, Germany